CLINICAL TRIAL: NCT01331473
Title: PROximal Protection VErsus NON-Protection in Carotid Artery Stenting (PROVENON Study) A Randomized Prospective MRI-based Trial.
Brief Title: PROximal Protection VErsus NON-Protection in Carotid Artery Stenting
Acronym: PROVENON
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Prof. Wolfgang Reith, Department of Diagnostic and Interventional Neuroradiology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROVENON01
Record Dates: First submitted 2011-03-30; First posted 2011-04-08 (Estimated); Last update posted 2011-12-05 (Estimated); Status verified 2011-03

CONDITIONS: Carotid Artery Stenosis
Keywords: Carotid Artery; Stenting; CAS; proximal protection
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carotid Artery Stenting without Protection (Active Comparator): Subjects will undergo carotid artery angioplasty and stenting with any CE-certificated carotid stent and without embolic protection device
  Interventions: Procedure: Carotid Artery Stenting without Protection
- Carotid Artery Stenting with Proximal Protection (Active Comparator): Subjects will undergo carotid artery angioplasty and stenting with any CE-certificated carotid stent and with a proximal embolic protection device provided by the GORE Neuro Protection System
  Interventions: Procedure: Carotid Artery Stenting with Proximal Protection

INTERVENTIONS:
Procedure: Carotid Artery Stenting with Proximal Protection — Carotid artery angioplasty and stenting with proximal embolic protection provided by the GORE Neuro Protection System
  Arms: Carotid Artery Stenting with Proximal Protection
Procedure: Carotid Artery Stenting without Protection — Carotid artery angioplasty and stenting without cerebral embolic protection
  Arms: Carotid Artery Stenting without Protection

SUMMARY:
To compare the incidence of new ischemic brain injury detected with magnetic resonance imaging (MRI) after carotid artery stenting in patients treated with and without proximal cerebral protection (Gore Flow Reversal System).

DETAILED DESCRIPTION:
Primary Objective:

The purpose of this study is to compare the rate of new ischemic brain injury detectable on MRI after carotid artery stenting between patients treated with proximal cerebral protection (Gore Flow Reversal System) and without cerebral protection.

Secondary Objective:

Impact of MRI-morphology of atherosclerotic plaque to the rate of new hyperintense diffusion weighted imaging (DWI) lesion on the post-treatment scan and to the rate of ipsilateral stroke or death.

ELIGIBILITY:
Inclusion Criteria:

* Male and female ≥ 18 years old;
* Suitable/Eligible for carotid artery revascularization;
* Significant artery stenosis in symptomatic patients defined as ≥ 50% of the artery diameter (%DS) or asymptomatic ≥ 80 %DS by angiography. Symptomatic is defined as a carotid artery stenosis associated with ipsilateral transient ischemic attack (TIA), amaurosis fugax, ischemic stroke or retinal infarction within 6 months prior to enrollment.
* Adequate clinical conditions to perform DW-MRI.
* Ability of the individual to understand the character and the consequences of clinical trial.
* Signed and dated informed consent provided before the beginning of any intervention.
* Negative pregnancy test (serum or urine) and contraception use for any woman of childbearing age. Systematic contraceptives (oral, implant, injection) and dia-phragm or condoms with spermicidal are considered reliable. Women who have undergone bilateral oophorectomy or/and hysterectomy or women status post-menopausal for at least two years are eligible for this trial.

Exclusion Criteria:

* Intracranial hemorrhage, hemorrhagic stroke, or stroke with mass effect demonstrated on CT scan or MRI within 30 days of the index procedure.
* Persisting ischemic stroke (defined as either a score > 15 on the NIH stroke scale, a Rankin score > 3 or a Barthel score < 60 measured within one week prior to study entry).
* Intracranial mass lesion (i.e., abscess, tumor, or other infection).
* peripheral vascular, supra-aortic or internal carotid artery tortuosity precluding the use of catheter-based techniques required for successful results.
* Lactation.
* Arterio-venous malformation in the territory of the target carotid artery.
* Any disease or medication that affects local hemostasis,
* Participation in other clinical trials during the present clinical trial or within the last month.
* Medical or psychological condition that would not permit completion of the trial or signing of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2011-05; Primary Completion 2014-05 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
The detection rate of new hyper-intense DWI lesion on the post-treatment compared to the pretreatment MRI imaging | Day 1-3

SECONDARY OUTCOMES:
Ipsilateral stroke (ischaemic stroke, intracerebral bleeding or both, with symptoms lasting more than 24 h) or death between treatment and 30 days after treatment | Day 30
Technical Success of the procedure | Day 0
  Subjects (both groups) who due to technical reaseons are unable to performe carotid artery stenting will be considered as technical failures.
  Subjects who are unable to tolerate flow reversal (in group 2) and have their procedures completed without embolic protection or other methods will be also considered as technical failures.
Access site vascular complications, defined as need for surgical repair or blood transfusion | Day 0-7

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Reith, MD, Principal Investigator — Saarland University Hospital
Locations (1):
- Department of Diagnostic and Interventional Neuroradiology, Homburg, Saarland, Germany

REFERENCES:
- [Background] Grunwald IQ, Papanagiotou P, Roth C, Fassbender K, Karp K, Krick C, Schieber H, Muller M, Haass A, Reith W. Lesion load in unprotected carotid artery stenting. Neuroradiology. 2009 May;51(5):313-7. doi: 10.1007/s00234-008-0491-6. Epub 2009 Feb 6. PMID 19198823
- [Background] Grunwald IQ, Papanagiotou P, Struffert T, Politi M, Krick C, Romaike BF, Ahlhelm F, Reith W. Reversal of flow during carotid artery stenting: use of the Parodi antiembolism system. Neuroradiology. 2007 Mar;49(3):237-41. doi: 10.1007/s00234-006-0178-9. Epub 2007 Jan 5. PMID 17205314
- [Background] Kastrup A, Nagele T, Groschel K, Schmidt F, Vogler E, Schulz J, Ernemann U. Incidence of new brain lesions after carotid stenting with and without cerebral protection. Stroke. 2006 Sep;37(9):2312-6. doi: 10.1161/01.STR.0000236492.86303.85. Epub 2006 Aug 3. PMID 16888277